CLINICAL TRIAL: NCT04367142
Title: Rapid Detection of COVID-19 by Portable and Connected Biosensor : Biological Proof of Concept
Brief Title: Rapid Detection of COVID-19 by Portable and Connected Biosensor
Acronym: COR-DIAL-1
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_36; 2020-A01147-32 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2023-05

CONDITIONS: Sars-CoV2
MeSH Terms: interventions — COVID-19 Nucleic Acid Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — nasopharyngeal swab and saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- positive SARS-Cov2: 100 patients with a positive diagnosis of SARS-CoV-2
  Interventions: Diagnostic Test: COVID-19 RT-PCR; Diagnostic Test: Biosensor
- negative SARS-Cov2: 100 patients with a negative diagnosis of SARS-CoV-2 defined by the gold standard by the medical team
  Interventions: Diagnostic Test: COVID-19 RT-PCR; Diagnostic Test: Biosensor

INTERVENTIONS:
Diagnostic Test: COVID-19 RT-PCR — Nasopharyngeal swabs for COVID-19 RT-PCR
Diagnostic Test: Biosensor — Portable and Connected Biosensor viral

SUMMARY:
The objective of study is to estimate the sensitivity and specificity of the COR-DIAL based on nasopharyngeal samples taken at the patient's admission in relation to the final diagnosis of COVID-19 made by the medical team.

ELIGIBILITY:
Inclusion Criteria:

* Male or female or child without age limit
* Admitted to a Reference Health Establishment in an emergency unit, hospitalisation or intensive care unit for suspicion of SARS-CoV-2 infection, regardless of the clinical presentation and degree of severity.
* Patient to be diagnosed using a PCR test on nasopharyngeal swab.
* Social insured

Exclusion Criteria:

* Atypical or suspicious cases without a final diagnosis of COVID-19 positive or negative
* Patient refusal to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients admitted to a Reference Health Establishment for suspicion of SARS-CoV-2
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the COR-DIAL based on nasopharyngeal swabs taken on admission of the patient compared to the final diagnosis of COVID-19 made by the medical team | Baseline (at admission)

SECONDARY OUTCOMES:
Cohen's Kappa Coefficient for concordance for the diagnosis of CoV-2-SARS between PCR and COR-DIAL based on nasopharyngeal swabs taken on patient admission | Baseline (at admission)

CONTACTS AND LOCATIONS:
Overall Officials: Enagnon Kazali ALIDJINOU, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHU lille, Lille, France